CLINICAL TRIAL: NCT02001636
Title: Impact of Protein Supplementation After Bariatric Surgery - a Randomized, Controlled, Double Blind Pilot Study
Brief Title: Effect of Protein Supplementation After Bariatric Surgery
Acronym: EPEAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Professor Dr. med. Stephan C. Bischoff, University of Hohenheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DONM-UHOH-386
Record Dates: First submitted 2013-11-20; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Protein Malnutrition
Keywords: Bariatric surgery; Protein malnutrition; Protein supplementation; Body composition; Body fat mass; Protein intake
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Protein group (Experimental): Patient group which takes daily protein supplements after bariatric surgery over 6 months.
  Protein product: Resource Instant Protein 88, Nestlé Health Nutrition
  Interventions: Drug: Resource Instant Protein 88
- Control group (Placebo Comparator): Patient group which takes daily isocaloric placebo after bariatric surgery over 6 months and thus can be compared to the protein group.
  Placebo product: Resource Maltodextrin, Nestlé Health Nutrition
  Interventions: Drug: Resource Maltodextrin

INTERVENTIONS:
Drug: Resource Instant Protein 88 — Protein product: Resource Instant Protein 88, Nestlé Health Nutrition; postoperative intake of 30 - 35 g powder per day over 6 months.
  Arms: Protein group
Drug: Resource Maltodextrin — Placebo product (Resource Maltodextrin, Nestlé Health Nutrition). Postoperative intake of 30 - 35 g powder per day over 6 months.
  Arms: Control group

SUMMARY:
Obese patients, who underwent bariatric surgery, are at risk to develop protein malnutrition. The aim of this study is to evaluate the influence of postoperative protein supplementation on weight reduction, body composition and protein status.

DETAILED DESCRIPTION:
Bariatric surgery has become a major treatment option for severe obesity in adults. It has proven its efficiency regarding weight loss and its benefits concerning the improvement or even remission of obesity related comorbidities. Additionally, bariatric surgery procedures can be performed laparoscopically, which decreases the complication rate and reduces postoperative pains. Despite the advantages of bariatric surgery, attention needs to be paid to the possible risks following the surgical treatment. Postoperative risks often concern the nutritional status. It has been shown that, beside different micronutrient deficiencies, bariatric surgery also leads to an increased risk of developing protein malnutrition. Discussed reasons for this are the malabsorption of nutrients and the restricted food intake after surgery, which may lead to reduced protein consumption. Postoperative occurrence of vomiting or different food intolerances may support this effect. Accordingly, if an inadequate supply persists, a protein deficit will occur and this, in turn, may lead to an undesirable reduction in muscle mass and plasma protein levels. Based on this background, numerous studies indicate an increased incidence of protein malnutrition after bariatric surgery by detecting a decrease in levels of albumin and prealbumin, a significant reduction in lean body mass, as well as an inadequate protein intake after surgical treatment.

Dietary proteins have shown to play an important role in body weight regulation. There is evidence that a protein-rich diet is supposed to facilitate weight loss, to support successful weight maintenance, to attain satiety and to preserve lean body mass. Therefore, the use of protein supplements after bariatric surgery may minimize the risk for developing protein malnutrition and hence optimize the postoperative care.

The primary aim of this randomized, placebo-controlled, double blind pilot study was to evaluate the influence of postoperative protein supplementation on body weight reduction, body composition and protein status.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* BMI of 35 kg/m2 or more
* Indication for laparoscopic sleeve gastrectomy or Roux-en Y gastric bypass

Exclusion Criteria:

* Renal disease
* Type 2 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Excess weight loss [%] | At month 6

SECONDARY OUTCOMES:
Content of lean body mass in lost weight [%] | At month 6
  Lean body mass is measured by using bioelectrical impedance analysis. The content of lean body mass in lost weight is calculated using the lost weight in kg and the lost lean body mass in kg.

OTHER OUTCOMES:
Content of body fat in lost weight [%] | At month 6
  Body fat mass is measured by using bioelectrical impedance analysis. The content of body fat mass in lost weight is calculated using the lost weight in kg and the lost body fat in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C Bischoff, Prof.Dr.med., Principal Investigator — Department of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany
Locations (1):
- Department of General, Visceral and Transplant Surgery, University Hospital of Tübingen, Tübingen, Germany